CLINICAL TRIAL: NCT00211445
Title: Photodynamic Therapy Using Verteporfin for Treatment of Chronic Central Serous Chorioretinopathy (CSC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT for CSC
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-09-28 (Estimated); Status verified 2007-09

CONDITIONS: Chronic Central Serous Chorioretinopathy
MeSH Terms: interventions — Photochemotherapy; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Photodynamic Therapy with Verteporfin
Drug: verteporfin

SUMMARY:
Central serous choroidal (CSC) retinopathy is a disease of the macula characterized by exudation of fluid under the retina localized to the posterior pole as well as loss of vision. The etiology is unknown, but according to the studies this condition is more common in young males and is associated with type A personality. Clinically, CSC is characterized by serous retinal detachment and area of leakage of in the subretinal space. The standard of care for acute CSC is observation for a period of up to 3 months. If there is no complete resolution of the retinal detachment by 3 months, there is an indication for focal laser photocoagulation therapy of the area of leakage. This treatment is usually effective in stopping leakage of fluid under the retina and causing resolution of detachment. However, laser photocoagulation therapy is not beneficial in the treatment of chronic CSC because there is not a single easily identifiable point of leakage but rather diffuse disease of RPE thus rendering laser treatment ineffective.The purpose of this medical research study is to evaluate Verteporfin therapy as an approach which may benefit patients with CSC, based on observations in exudative type of AMD patients treated with Photodynamic Therapy using Verteporfin.

DETAILED DESCRIPTION:
7.1 Visit 1 - Screening Visit

The first visit by the patient is for the purpose of screening the patient for the study. This visit must occur within 1 week prior to the treatment visit. At this visit the investigator and the supporting staff will:

1. Determine if the patient is eligible for enrollment in the study, explain the study to the patient, and obtain an informed consent from the patient. The form should be witnessed and documented by obtaining the patient's signature at this visit.
2. Only one eye of the patient can be enrolled in the study. For patients with lesions in both eyes, the investigator may enroll the eye they deem most eligible or amenable to treatment.
3. Record patient demographics, complete medical history and contact information on the initial visit form.
4. Perform a complete eye examination including:

   i. visual acuity. ii. slit-lamp biomicroscopy. iii. dilated fundus examination.
5. Obtain stereo color fundus photographs (30 degree field of view) of the study eye.
6. Obtain sodium fluorescein angiogram of the study eye via digital imaging system.
7. Obtain ICGA of the study eye. NOTE: If a patient presents with any acute illness during screening and the day of treatment administration, his entry into the study is deferred until the acute illness resolves.

7.2 Visit 2 - Treatment Visit (Day Zero)

At this visit the patient is assigned a Verteporfin-PDT laser energy delivery profile according to the scheme detailed in Section 5.1, above. The investigator and the supporting staff will:

1. Perform an eye examination including best-corrected visual acuity using the EDTRS visual chart.
2. The angiograms may need to be repeated if the previous angiograms were done more than 72 hours ago.
3. Perform Verteporfin-PDT treatment. NOTE: If a patient presents with any acute illness during screening and the day of treatment administration, his entry into the study is deferred till the acute illness resolves.

7.3 Visit 3 & 4- First Post-treatment Follow-up Visit

The investigator will have the patient return to the office after 2 weeks (Visit 3) and 6 weeks (Visit 4) after performing the Verteporfin-PDT treatment. At this visit the investigator and the supporting staff will:

1. Perform a complete eye examination including

   1. best corrected visual acuity using EDTRS visual acuity chart.
   2. slit-lamp biomicroscopy.
   3. dilated fundus examination.
2. Obtain stereo color fundus photographs (30 degree field of view) of the study eye.
3. Obtain sodium fluorescein angiogram of the study eye via digital imaging system.
4. Obtain ICGA of the study eye.
5. Ask the patient about any new ocular or systemic symptoms that developed since last visit, and look for any associated signs and record both on the case report forms.
6. Ask the patient and record any new medications being used since the last visit.
7. If the patient is re-treated then the post-treatment visit schedule will start again at visit 3 as detailed in Section 7.3 Visit 3.

7.4 Visit 5 through Visit 12 - Follow-up Visits

The investigator will have the patient return to the office at 3-month (plus/minus 2 weeks) intervals after performing the last Verteporfin-PDT treatment. The visit windows are continuous, but two consecutive visits should not be scheduled within 2 weeks of each other. At these visits the investigator and the supporting staff will:

1. Perform a complete eye examination including

   1. best corrected visual acuity using EDTRS visual acuity chart.
   2. slit lamp biomicroscopy.
   3. dilated fundus examination.
2. Obtain stereo color fundus photographs (30 degree field of view) of the study eye.
3. Obtain sodium fluorescein angiogram of the study eye.
4. Obtain ICGA of the study eye.
5. Ask the patient about any ocular or systemic symptoms, and look for any associated signs and record both on the case report forms.
6. Ask the patient and record any medications being used.
7. Based on the eye examination and the ICGA the investigator must decide whether any new or previously treated CNV vessels need to be treated.
8. Perform any additional or concomitant treatment as required.
9. At the final visit (approximately 24 months after entry into the study), the patient will be terminated from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of chronic central serous chorioretinopathy and clinical/angiographic findings typical of the disease of greater than 6 months duration.Chronic central serous chorioretinopathy could be defined on the basis of two factors: a) persistence of the detachment for more than 6 months and b) chronic recurrent acute detachments with widespread decompensation of the retinal pigment epithelium.
2. VA 20/40 and 20/320 Study Eye on the ETDRS visual acuity chart.
3. VA 20/800 or better Fellow Eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with tears in retinal pigment epithelium.
2. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
3. Patients who have undergone intraocular surgery within last 2 months or capsulotomy within last month in study eye.
4. Patient participating in any other investigational drug study.
5. Inability to obtain photographs to document CNV (including difficulty with venous access).
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to indocyanine green or iodine.
8. Patient is pregnant or nursing
9. Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-07; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
mean change in VA (ETDRS) from baseline to 24 months | 24 months
investigate the potential of photodynamic therapy using verteporpin in chronic central serous chorioretinopathy | 24 months

SECONDARY OUTCOMES:
mean change of VA(ETDRS), OCT, FA from baseline to 24 months | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason S. Slakter, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States